CLINICAL TRIAL: NCT03383380
Title: Efficacy and Safety of Rapamycin Therapy for Patients With Activated Phosphoinositide 3-Kinase δ Syndrome
Brief Title: Rapamycin Treatment for Activated Phosphoinositide 3-Kinase δ Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Jinqiao Sun, Professor, Children's Hospital of Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTAPDS
Record Dates: First submitted 2017-12-12; First posted 2017-12-26 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Activated PI3K-delta Syndrome; Immunodeficiency Primary
Keywords: Activated PI3K-delta Syndrome; Immunodeficiency Primary; Akt/mTOR pathway; Rapamycin Therapy; Hyperphosphorylation
MeSH Terms: conditions — Activated PI3K-delta Syndrome; Primary Immunodeficiency Diseases | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rapamycin (Experimental): Treatment for patients with activated phosphoinositide 3-kinase δ syndrome
  Interventions: Drug: Rapamycin

INTERVENTIONS:
Drug: Rapamycin — Gain-of-function (GOF) PIK3CD mutations lead to PI3Kδ hyperactivity, with the downstream mediators Akt and mTOR hyperphosphorylated. The mammalian/mechanistic target of rapamycin inhibitor rapamycin may be effective to control the progress of this disease.
  Other Names: Sirolimus

SUMMARY:
The purpose of this proposed research is to evaluate the efficacy and safety of the rapamycin therapy in patients with activated phosphoinositide 3-kinase δ syndrome (APDS).

DETAILED DESCRIPTION:
Activated phosphoinositide 3-kinase δ syndrome (APDS) is a recently described autosomal dominant primary immunodeficiency (PID), caused by the mutations in PIK3CD gene. The manifestations of APDS mainly include recurrent respiratory tract infections, persistent Epstein-Barr virus (EBV)/ cytomegalovirus (CMV)infections, lymphadenopathy, splenomegaly, CD4+T cells lymphopenia, and hyper-IgM syndrome. PIK3CD encodes p110δ, the catalytic subunit of phosphatidylinositol 3-kinase (PI3K) which mainly expresses in leukocytes, being critical for their proliferation, activation and survival. Gain-of-function (GOF) PIK3CD mutations lead to PI3Kδ hyperactivity, with the downstream mediators Akt and mammilian target of rapamycin (mTOR) hyperphosphorylated. Patient-derived lymphocytes had increased levels of phosphatidylinositol 3,4,5-trisphosphate and phosphorylated AKT protein. Hyperactivation of mTOR increases phosphorylation of kinases and increased glycolysis that results in enhanced proliferation and senescence of terminally differentiated CD8+ Tcell populations.

The optimal treatment for these APDS patients is not yet determined; however, there are many kinds of therapeutic approaches (anti-infection prophylaxis, immunoglobulin replacement, conventional immunosuppressants, PI3K/mTOR inhibitors and hematopoietic stem cell transplantation). The APDS patients frequently receive treatment with immunoglobulin replacement and antibiotics. Hematopoietic stem cell transplantation (HSCT) has been currently curative in APDS patients; however, longer-term follow-up to determine the degree of donor chimerism and efficacy is required. There are several subjects without a prompt suitable matched donor or for whom the critical disease conditions force to postpone HSCT.The mammalian/mechanistic target of inhibitor rapamycin was reported to improve circulating T-cell profiles. Individual patients in previous studies experienced a decrease in nonneoplastic lymphoproliferation while taking rapamycin.

The investigators in this study hope to evaluate the efficacy and safety of rapamycin in the treatment for carefully selected patients with APDS.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with activated phosphoinositide 3-kinase δ syndrome
2. No more than 18 years old

Exclusion Criteria:

1. Patients with serious fungous infection
2. Patients with serious complications
3. Lack of parental consent

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Frequency of Recurrent Infections | 5 years
  Frequency of recurrent infections of the patients as indicators of rapamycin efficacy.
Hepatosplenomegaly | 5 years
  Changes in hepatosplenomegaly with rapamycin treatment.
Lymphocyte subset | 5 years
  The changes of lymphocytes subset were evaluated by flow cytometry.

SECONDARY OUTCOMES:
Incidence of Adverse Events | 5 years
  Unexpected toxic adverse events during and after using rapamycin

CONTACTS AND LOCATIONS:
Overall Officials: Jinqiao Sun, Ph.D.,M.D, Principal Investigator — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coulter TI, Chandra A, Bacon CM, Babar J, Curtis J, Screaton N, Goodlad JR, Farmer G, Steele CL, Leahy TR, Doffinger R, Baxendale H, Bernatoniene J, Edgar JD, Longhurst HJ, Ehl S, Speckmann C, Grimbacher B, Sediva A, Milota T, Faust SN, Williams AP, Hayman G, Kucuk ZY, Hague R, French P, Brooker R, Forsyth P, Herriot R, Cancrini C, Palma P, Ariganello P, Conlon N, Feighery C, Gavin PJ, Jones A, Imai K, Ibrahim MA, Markelj G, Abinun M, Rieux-Laucat F, Latour S, Pellier I, Fischer A, Touzot F, Casanova JL, Durandy A, Burns SO, Savic S, Kumararatne DS, Moshous D, Kracker S, Vanhaesebroeck B, Okkenhaug K, Picard C, Nejentsev S, Condliffe AM, Cant AJ. Clinical spectrum and features of activated phosphoinositide 3-kinase delta syndrome: A large patient cohort study. J Allergy Clin Immunol. 2017 Feb;139(2):597-606.e4. doi: 10.1016/j.jaci.2016.06.021. Epub 2016 Jul 16. PMID 27555459
- [Background] Lucas CL, Kuehn HS, Zhao F, Niemela JE, Deenick EK, Palendira U, Avery DT, Moens L, Cannons JL, Biancalana M, Stoddard J, Ouyang W, Frucht DM, Rao VK, Atkinson TP, Agharahimi A, Hussey AA, Folio LR, Olivier KN, Fleisher TA, Pittaluga S, Holland SM, Cohen JI, Oliveira JB, Tangye SG, Schwartzberg PL, Lenardo MJ, Uzel G. Dominant-activating germline mutations in the gene encoding the PI(3)K catalytic subunit p110delta result in T cell senescence and human immunodeficiency. Nat Immunol. 2014 Jan;15(1):88-97. doi: 10.1038/ni.2771. Epub 2013 Oct 28. PMID 24165795
- [Background] Tsujita Y, Mitsui-Sekinaka K, Imai K, Yeh TW, Mitsuiki N, Asano T, Ohnishi H, Kato Z, Sekinaka Y, Zaha K, Kato T, Okano T, Takashima T, Kobayashi K, Kimura M, Kunitsu T, Maruo Y, Kanegane H, Takagi M, Yoshida K, Okuno Y, Muramatsu H, Shiraishi Y, Chiba K, Tanaka H, Miyano S, Kojima S, Ogawa S, Ohara O, Okada S, Kobayashi M, Morio T, Nonoyama S. Phosphatase and tensin homolog (PTEN) mutation can cause activated phosphatidylinositol 3-kinase delta syndrome-like immunodeficiency. J Allergy Clin Immunol. 2016 Dec;138(6):1672-1680.e10. doi: 10.1016/j.jaci.2016.03.055. Epub 2016 Jul 14. PMID 27426521
- [Background] Vignesh P, Rawat A, Singh S. An Update on the Use of Immunomodulators in Primary Immunodeficiencies. Clin Rev Allergy Immunol. 2017 Apr;52(2):287-303. doi: 10.1007/s12016-016-8591-2. PMID 27873163
- [Background] Angulo I, Vadas O, Garcon F, Banham-Hall E, Plagnol V, Leahy TR, Baxendale H, Coulter T, Curtis J, Wu C, Blake-Palmer K, Perisic O, Smyth D, Maes M, Fiddler C, Juss J, Cilliers D, Markelj G, Chandra A, Farmer G, Kielkowska A, Clark J, Kracker S, Debre M, Picard C, Pellier I, Jabado N, Morris JA, Barcenas-Morales G, Fischer A, Stephens L, Hawkins P, Barrett JC, Abinun M, Clatworthy M, Durandy A, Doffinger R, Chilvers ER, Cant AJ, Kumararatne D, Okkenhaug K, Williams RL, Condliffe A, Nejentsev S. Phosphoinositide 3-kinase delta gene mutation predisposes to respiratory infection and airway damage. Science. 2013 Nov 15;342(6160):866-71. doi: 10.1126/science.1243292. Epub 2013 Oct 17. PMID 24136356
- [Background] Walsh CM, Fruman DA. Too much of a good thing: immunodeficiency due to hyperactive PI3K signaling. J Clin Invest. 2014 Sep;124(9):3688-90. doi: 10.1172/JCI77198. Epub 2014 Aug 18. PMID 25133419